CLINICAL TRIAL: NCT05296564
Title: A Phase I/II Dose Escalation, Safety and Efficacy Study of Anti-NY-ESO-1 T Cell Receptor (TCR)-Gene Engineered Lymphocytes Given by Infusion to Patients With NY-ESO-1 -Expressing Metastatic Cancers
Brief Title: Anti-NY-ESO-1 TCR-Gene Engineered Lymphocytes Given by Infusion to Patients With NY-ESO-1 -Expressing Metastatic Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0752-20-HMO
Record Dates: First submitted 2022-02-22; First posted 2022-03-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Sarcoma, Synovial; Sarcoma,Soft Tissue; Melanoma Stage IV; Triple Negative Breast Cancer; Metastatic Cancer; Non Small Cell Lung Cancer; Bladder Urothelial Carcinoma; Neuroblastoma, Metastatic; Ovary Cancer
Keywords: NY-ESO-1; TCR; adoptive transfer; retroviral transduction
MeSH Terms: conditions — Sarcoma, Synovial; Sarcoma; Melanoma; Triple Negative Breast Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Neuroblastoma; Ovarian Neoplasms | interventions — Cyclophosphamide; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HBI 0201-ESO TCRT (Anti-NY-ESO-1 TCR-transduced peripheral blood lymphocytes) (Experimental): This is a two-part, non-randomized, open label, single-site Phase I/II study. The first Part A is a dose ranging maximum tolerated dose (MTD) study and Part B is an extension phase to evaluate safety at the selected safe dose. A Data Safety Monitoring Board (DSMB) will determine the safe dose for testing in the expansion phase (Part B).
  Part A will be according to a 3+3 dose escalation design. A total of up to 20 patients will participate in this Part.
  Part B will be an expansion phase. The objective will be to determine if the treatment regimen is associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% Partial Response (PR) + Complete Response (CR) rate (p1=0.20).
  A total of up to 43 patients may be enrolled in Part B (41 +2, allowing for up to 2 non-evaluable patients).
  Interventions: Drug: CYCLOPHOSPHAMIDE and FLUDARABIN; Drug: Cyclophosphamide; Biological: HBI 0201-ESO TCRT; Drug: Aldesleukin

INTERVENTIONS:
Drug: CYCLOPHOSPHAMIDE and FLUDARABIN — 1. CYCLOPHOSPHAMIDE 250 mg/msq, Day -5,-4,-3 with FLUDARABIN 25 mg/msq, Day -5,-4,-3
  Other Names: CYTOXAN
Drug: Cyclophosphamide — CYCLOPHOSPHAMIDE 250 mg/msq, Day -6, -5,-4,-3
  Other Names: CYTOXAN
Biological: HBI 0201-ESO TCRT — HBI 0201-ESO TCRT will be infused on Day 0, after lymphodepletion. Three dose levels will be evaluated: 1x10E9, 5x10E9 and 1x10E10.
Drug: Aldesleukin — Continuous infusion of aldesleukin 18x10E6 IU/24h will be given 24 hours post HBI 0201-ESO TCRT infusion, for four days or until a dose limiting toxicity will occur that mimics cytokine release syndrome (CRS) including blood pressure drop, oliguria or confusion- all of them or any one alone.
  Other Names: Interleukin-2

SUMMARY:
A Phase I/II Dose Escalation, Safety and Efficacy Study of HBI 0201-ESO TCRT (anti-NY-ESO-1 TCR-Gene Engineered Lymphocytes) Given by Infusion to Patients with NY-ESO-1 -Expressing Metastatic Cancers

DETAILED DESCRIPTION:
This is a two-part, non-randomized, open label, single-site Phase I/II study. The first Part A is a dose ranging maximum tolerated dose (MTD) study and Part B is an extension phase to evaluate safety at the selected safe dose. A Data Safety Monitoring Board (DSMB) will determine the safe dose for testing in the expansion phase (Part B).

Part A will be according to a 3+3 dose escalation design. A total of up to 20 patients will participate in this Part.

Part B will be an expansion phase. The objective will be to determine if the treatment regimen is associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% Partial Response (PR) + Complete Response (CR) rate (p1=0.20).

A total of up to 43 patients may be enrolled in Part B (41 +2, allowing for up to 2 non-evaluable patients).

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed diagnosis of neoplasia
2. Measurable (per RECIST v1.1 criteria) metastatic cancer or locally advanced refractory/recurrent malignancy not amenable to curative treatment. Lesions previously irradiated may be considered measurable only if growth has been documented since local treatment completion.
3. The tumor expresses ESO as assessed immunohistochemistry of resected tissue. To this end, archived tumor tissue suitable for analysis must be available or re-biopsy performed on study. Tissue staining must encompass more than 10% of tumor section.
4. Patients must have previously either (1) received at least first-line or second-line standard therapy for metastatic disease, if known to be effective for that disease, and have been either non-responders (progressive disease), intolerable or have recurred or (2) Recurred within 6 months of adjuvant systemic therapy known to be active also in the metastatic setting.
5. Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
6. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
7. Age ≥ 18 years and ≤ 70 years.
8. Patient is able to understand and willing to sign a written informed consent.
9. Clinical performance status of ECOG 0, 1 or 2.
10. HLA-A*0201or A*0206 positive.
11. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for four months after treatment.
12. Women of child-bearing potential must have a negative pregnancy test.
13. Serology: Seronegative for HIV antibody, hepatitis B antigen, and hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
14. Hematology

    * ANC > 1500/mm3 without the support of filgrastim
    * WBC ≥ 3000/mm3
    * Platelet count ≥ 100,000/mm3
    * Hemoglobin > 8.0 g/dL. Subjects may be transfused to reach this cut-off.
15. Chemistry

    * Serum ALT/AST ≤ 2.5 x ULN
    * Creatinine clearance ≥40ml/min
    * Total bilirubin ≤ 1.5 mg/dL, except in patients with Gilbert's Syndrome, who must have a total bilirubin < 3.0 mg/dL.
    * INR < 1.5

Exclusion Criteria:

1. Women of child-bearing potential who are pregnant or breastfeeding.
2. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
3. Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses
4. Concurrent systemic steroid therapy, not including replacement therapy or treatment with prednisone up to 10mg daily or its equivalent. Or any other form of immunosuppressive therapy within 7 days before the first dose of study intervention.
5. History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
6. Subjects with a history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within 3 months.
7. Subjects unable to maintain normal oxygen saturation level in room air.
8. Subjects who have had a venous thromboembolic event requiring anticoagulation and who meet any of the following criteria:

   * Have been on a stable dose of anticoagulation for < 1 month (except for acute line insertion induced thrombosis).
   * Have had a Grade 2, 3, or 4 hemorrhage in the last 30 days or are experiencing continued symptoms from their venous thromboembolic event (e.g. continued dyspnea or oxygen requirement).
9. Has a known additional malignancy within the last 3 years. Exceptions include early stage cancers (carcinoma in situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy).
10. LVEF ≤ 40%
11. Documented FEV1 ≤ 60% predicted tested in patients with:

    * A prolonged history of cigarette smoking (≥ 20 pack-year smoking history, with cessation within the past two years).
    * Symptoms of respiratory dysfunction.
12. Patients who are at the time of study initiation receiving any other investigational agents.
13. Carcinomatosis meningitis or other brain involvement exceeding that allowed above.
14. Has received live vaccine within 30 days before the first dose of study intervention. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 5 years
  Adverse events that occur following engineered T cell transfer
objective tumor regression | 5 years
  change in index lesions' size

SECONDARY OUTCOMES:
immune monitoring for transferred cells persistence | 5 years
  blood test for ESO-TCRT cells' presence

CONTACTS AND LOCATIONS:
Overall Officials: Michal Lotem, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No